CLINICAL TRIAL: NCT07075172
Title: Instrument Assisted Soft Tissue Mobilization Alters the Material and Mechanical Properties of Healthy, Shortened Achilles Tendons: a Within-subject Randomized Controlled Study
Brief Title: Does Instrument-assisted Mobilization Influence Healthy, Short Achilles Tendons?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Stuart Warden, Professor of Physical therapy, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BaylissRCT1
Record Dates: First submitted 2025-06-18; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Achilles Tendon Length and Thickness

STUDY DESIGN:
Intervention Model Description: Within-subject controlled study. One side of the body is treated with the other side being an internal non-treated control site.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IASTM treated (Experimental): Leg treated with instrument-assisted soft tissue mobilization
  Interventions: Other: Instrumented-assisted soft tissue mobilization
- Non-treated (No Intervention): Non-treated leg

INTERVENTIONS:
Other: Instrumented-assisted soft tissue mobilization — Instrumented-assisted soft tissue mobilization of the posterior leg and Achilles tendon region
  Arms: IASTM treated

SUMMARY:
The goal of this clinical trial is to learn if instrumented-assisted soft tissue mobilization (i.e., massage using specialized metal instruments) of the lower leg and Achilles tendon region changes the properties of the tendon and the range of ankle dorsiflexion (i.e., the ability to bring the foot and toes back towards the head).

One lower leg and Achilles tendon in each participant will be treated with instrumented-assisted soft tissue mobilization for 7 minutes during 8 treatment sessions over a 4-week period. The other lower leg and Achilles tendon will not be treated and be assessed as the non-treated control leg.

DETAILED DESCRIPTION:
Tendons play a critical role in transferring muscle-generated forces to the skeleton for locomotion, but they are not solely force conveyors. Tendons also function as both mechanical buffers and power amplifiers. In their buffering role, tendons delay and slow muscle fascicle lengthening to dissipate energy during rapid negative work (i.e. eccentric contractions). However, it is in their role as power amplifiers that tendons have received most attention. Acting in a spring-like manner, tendons store elastic strain energy when stretched and return it when released to reduce the energy cost of motion. The amount of energy stored depends on a tendon's mechanical properties and, in particular, its stiffness.

Stiffness represents the ability of a structure to resist deformation and is dependent upon both the quality of material present (i.e. amount and type) and how it is arranged (i.e. structure). Stiffer tendons may promote an improved ability to transmit muscle-generated forces resulting in improved performance. A stiffer tendon may also protect against injury. Tendons experience failure in a relatively set strain (i.e. elongation) range. A stiffer tendon experiences less strain per unit of applied force and, thus, can withstand greater load before reaching damage-inducing strains.

It is now accepted tendons adapt their stiffness (among other properties) to their environment. Tendon stiffness declines with disuse, pathology (i.e. tendinopathy) and aging. Conversely, systematic reviews have demonstrated tendon stiffness increases in response to heightened levels of physical activity, with a preference toward high intensity loads (i.e. >70% maximum voluntary contraction or repetition maximum). However, beyond physical activity there are limited clinically available modalities to positively influence tendon stiffness. For instance, vibration and stretching interventions have not been shown to impact tendon stiffness or even cause it to decline.

A modality that may modulate tendon stiffness is instrument assisted soft tissue mobilization (IASTM). IASTM is a popular alternative to traditional manual therapy techniques and involves the use of specialized hard tools to apply controlled, localized mechanical loads to soft connective tissues. Initial preclinical animal studies reported IASTM altered fibroblast recruitment and activation after chemically-induced tendon injury, and improved tissue perfusion and mechanical recovery following surgically-induced ligament injury. Clinically, there is emerging but limited and low-quality evidence of the efficacy of IASTM in improving range of motion, pain and patient-reported outcomes. With regards to tissue stiffness, studies have reported single IASTM treatments targeting muscle to have no effect on musculotendinous shear modulus or stiffness, and to reduce or have no effect on passively assessed joint stiffness. To our knowledge, no study has reported a beneficial effect of IASTM on tendon mechanical and material properties, with Ikeda et al. reporting that IASTM self-administered over 6-weeks to the posterior lower leg had no impact on Achilles tendon (AT) shear modulus assessed using shear wave elastography.

The primary aim of the current study is to explore the effect of IASTM administered to the posterior lower leg and Achilles tendon twice per week for 4 weeks on the material and mechanical properties of the tendon in healthy subjects with reduced tendon length. A secondary aim is to investigate the impact of IASTM applied to the AT on range of ankle dorsiflexion, assessed using the weight bearing lunge ('lunge') test. The study will implement a within-subject controlled design wherein one leg received IASTM and the contralateral leg served as a non-IASTM treated internal control. Both sides will be equally exposed to warm-up and stretching activities within each treatment session.

ELIGIBILITY:
Inclusion Criteria:

* The distance from the tip of the great toe to the wall during the weightbearing lunge test is <90 mm bilaterally with ≤15 mm asymmetry
* A stretch sensation is reported in the region of the Achilles tendon during the weightbearing lunge test

Exclusion Criteria:

* A history of Achilles tendon injury, pain, rupture or surgery
* Current pain in the heel, foot or ankle
* Surgery in the past 12 months to the foot, heel or ankle
* A sensation other than a stretch within the Achilles tendon region during the weightbearing lunge test (e.g. compression/pinching in the vicinity of the anterior talocrural joint or a more vague, deeper stretch within the vicinity of the posterior talocrural joint).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-10-03 (Actual); Primary Completion 2014-10-16 (Actual); Study Completion 2014-10-16 (Actual)

PRIMARY OUTCOMES:
Change in the stiffness of the Achilles tendon measured using ultrasound | From enrollment until 6 days after the end of treatment at 4 weeks
  Participants will push their foot against a force measuring platform. At the same time, an ultrasound will be used to image their Achilles tendon. How much force they generated will be divided by how far the tendon stretches to indicate stiffness in newtons per millimeter (N/mm)
Change in the modulus of the Achilles tendon measured using ultrasound | From enrollment until 6 days after the end of treatment at 4 weeks
  Participants will push their foot against a force measuring platform. At the same time, an ultrasound will be used to image their Achilles tendon. How much force they generated will be divided by how far the tendon stretches to indicate stiffness in newtons per millimeter (N/mm). The stiffness will be divided by the cross sectional area of the tendon to indicate modulus in megaPascals (MPa).

SECONDARY OUTCOMES:
Range of motion of ankle dorsiflexion | From enrollment until 6 days after the end of treatment at 4 weeks
  Assessed using the weightbearing lunge test

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Warden, Principal Investigator — Indiana University Indianapolis
Locations (1):
- Indiana University Indianapolis, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be available from the study investigators upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months after the publication of results with no end date.
Access Criteria: Individuals can contact the investigators in writing to complete a data use agreement. Once approved by an institutional signing official, individual participant data will be provided.